CLINICAL TRIAL: NCT07143123
Title: An Action Research on Improving Clinical Nursing Skills of Nursing Students by Intervening With the SimCapture Cloud Management System
Brief Title: Enhancing Nursing Skills With SimCapture Technology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMUH113-REC2-058
Record Dates: First submitted 2025-04-28; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Motivation; Clinical Skills Training; Nursing Students; OSCE (Objective Structured Clinical Examination)

STUDY DESIGN:
Intervention Model Description: 1. The SimCapture system is used as a platform for managing, recording, and evaluating student learning.
  2. Both teachers and students have individual accounts to access the system.
  3. Teachers create digital evaluation tools for each skill.
  4. Students record their practice sessions and upload the videos to the SimCapture cloud.
  5. Teachers use tablets to provide feedback on student performance within the system.
  6. Students can review their own videos, as well as those of their peers, along with teacher feedback.
  7. SimCapture is used both within the skills lab and remotely, allowing students to practice and review independently.
  8. The system also allows for learning portfolios to track student progress.
Masking Description: No additional parties were masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SimCapture-Based Nursing Skills Training (Experimental)
  Interventions: Behavioral: Cloud-based learning platform

INTERVENTIONS:
Behavioral: Cloud-based learning platform — The SimCapture system is the technological backbone of the intervention, transforming the way clinical skills are taught and learned.
  1. System Access and Structure:Both faculty and students are provided with individual accounts to access the SimCapture platform.
  2. The system facilitates the organization of students into groups, enabling collaborative learning and peer feedback.
  3. Digital Evaluation Tools:Faculty develop standardized, digital tools within SimCapture to assess student performance of clinical skills.These tools ensure consistent and objective evaluation.
  4. Recording and Feedback:Students record their practice sessions using personal devices (e.g., smartphones).These recordings are uploaded to the SimCapture cloud, creating a repository of learning resources.
  5. Faculty use tablets to provide specific, time-stamped feedback on student performance directly within the SimCapture system.

SUMMARY:
The action research aims to enhance clinical nursing skills of nursing students through the implementation of the SimCapture cloud management system. Research has found that traditional teaching methods are insufficient in cultivating students' clinical skills, and students' learning characteristics and technological developments have also placed new demands on teaching. Although the research team previously attempted blended learning and simulation-based teaching, students' technical grades have shown a declining trend. To address this issue, the researchers plan to implement the SimCapture system and, based on observational learning theory, design teaching activities to enhance students' learning motivation and self-efficacy, ultimately improving their clinical skills.

ELIGIBILITY:
Inclusion Criteria:

１．Undergraduate nursing students in the 2nd or 3rd year

２．Enrolled in the applicant's clinical skills course during the academic year

Exclusion Criteria:

１．Students who have previously attempted and failed this course and are required to retake it

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
OSCE (Objective Structured Clinical Examination) Scores | At week 8 (mid-semester) and at week 16 (end of semester)
  The OSCE content includes preparation of technical equipment and technical procedures, which will be evaluated using a checklist by examiners.
  The checklist has undergone validity analysis by five nursing experts. Scores range from 0 to 100.

SECONDARY OUTCOMES:
Self-Efficacy Questionnaire | Weekly at weeks 1-17 of semester, within 3 days after each class
  This study developed a self-efficacy scale for technical courses based on Bandura's (1986) self-efficacy theory, which includes three dimensions: level, generality, and strength. Considering the potential burden on students from completing multiple items, the scale consists of three items: (1) "If I try my best, I can always complete the technical task"; (2) "With my abilities, I can handle even the most difficult or complex technical tasks"; and (3) "When facing challenges in learning technical skills, I can usually find several ways to overcome them." Higher scores indicate greater self-efficacy. The content validity of the questionnaire will be reviewed and revised through expert evaluation.
Learning Motivation Questionnaire | At week 1 (beginning of semester), week 9 (after midterm exam), and week 18 (final exam)]
  This study adopted a revised version of the Learning Motivation Scale (LMS) developed by Liu Cheng-Hung (2010) in Taiwan. The scale was adapted from the Motivated Strategies for Learning Questionnaire (MSLQ) by Pintrich, Smith, Garcia, and McKeachie (1991), taking into account the Taiwanese cultural context. The scale consists of 14 items and is one of the most widely used instruments for assessing learning motivation. Higher scores indicate stronger learning motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
We will share the anonymized individual participant data from this study to facilitate future research. The shared dataset will include demographic data (age, gender, ethnicity), baseline characteristics (disease severity, medical history), treatment data (drug dosage, duration), and primary outcome measurements (symptom scores, quality of life). Direct identifiers such as names, addresses, and dates of birth have been removed. The data will be made available through a secure online database, and a data access agreement will be required to access the data. The data will be available 12 months after the publication of the study and will be retained for 5 years.
  By providing a comprehensive and transparent description of the specific IPD to be shared, you can promote responsible data sharing and maximize the impact of the research, while protecting the privacy of participants.

REFERENCES:
- [Result] Nursing A, Council M. National competency standards for the registered nurse: Australian Nursing and Midwifery Council; 2005. Zieber M, Sedgewick M. Competence, confidence and knowledge retention in undergraduate nursing students-A mixed method study. Nurse Education Today. 2018;62:16-21. Waxman K. The development of evidence-based clinical simulation scenarios: guidelines for nurse educators. Journal of nursing education. 2010;49(1):29-35. Leidl DM, Ritchie L, Moslemi N. Blended learning in undergraduate nursing education-A scoping review. Nurse Education Today. 2020;86:104318. simulations in nurse education: A systematic mapping review. Nurse education today. 2021;101:104868. Bandura A. Social foundations of thought and action. Englewood Cliffs, NJ. 1986;1986(23-28). Catania A. Learning (interim 4th ed.). Cornwall-on-Hudson, NY: Sloan. 2007. 13. Devi B, Khandelwal B, Das M. Application of Bandura's social cognitive theory in the technology enhanced, blended learning environment. International Journal of Applied Research. 2017;3(1):721-724. Strand I, Gulbrandsen L, Slettebø Å, Nåden D. Digital recording as a teaching and learning method in the skills laboratory. Journal of clinical nursing. 2017;26(17-18):2572-2582. Stone R, Cooke M, Mitchell M. Undergraduate nursing students' use of video technology in developing confidence in clinical skills for practice: A systematic integrative literature review. Nurse Education Today. 2020/01/01/ 2020;84:104230. Bandura A, Grusec JE, Menlove FL. Observational learning as a function of symbolization and incentive set. Child development. 1966:499-506. Bandura A, Jeffrey RW. Role of symbolic coding and rehearsal processes in observational learning. Journal of personality and social psychology. 1973;26(1):122. 19. Huun KM. Directed observational learning through augmented video s

DOCUMENTS (1):
  • Study Protocol (2025-08-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT07143123/Prot_000.pdf